CLINICAL TRIAL: NCT04211064
Title: Comparison Of The Effects Of Deep And Moderate Neuromuscular Blockade On Optic Nerve Sheath Diameter İn Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Comparison of the Effects of Deep and Moderate Neuromuscular Blockade on Optic Nerve Sheath Diameter
Acronym: MBLONDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Serdar Yeşiltaş, Principle Investigator, Medical Doctor, Anesthesiology and Reanimation, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 54022451-050.05.04-
Record Dates: First submitted 2019-12-04; First posted 2019-12-26 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Intracranial Hypertension
Keywords: optic nerve sheath diameter; deep neuromuscular block; moderate neuromuscular block; intracranial hypertension
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into 2 groups. In the first group (Group 1), patients undergoing intraabdominal insufflation pressure 12 mmHg and deep neuromuscular block (TOF -- PTC 1-5), in the second group (Group 2) patients undergoing intraabdominal insufflation pressure 12 mmHg and moderate neuromuscular block (TOF 1-3) It would be classified.
Who Masked: Participant, Investigator
Masking Description: The participants were blinded to group allocation, as the measurements were performed after induction of general anesthesia. The investigator measuring the optic nerve sheath diameter was blinded to the group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep neuromuscular block (Other): Patients undergoing deep neuromuscular blockade with rocuronium (TOF -- PTC 1-5)
  Interventions: Diagnostic Test: Ultrasonographic measurement of optic nerve sheath diameter; Procedure: Deep neuromuscular block
- Moderate neuromuscular block (Active Comparator): Patients undergoing moderate neuromuscular blockade with rocuronium (TOF 1-3)
  Interventions: Diagnostic Test: Ultrasonographic measurement of optic nerve sheath diameter; Procedure: Moderate neuromuscular block

INTERVENTIONS:
Diagnostic Test: Ultrasonographic measurement of optic nerve sheath diameter — Optic nerve sheath diameter will be measured at both neuromuscular blocks level.
Procedure: Deep neuromuscular block — Deep neuromuscular block will be obtained via appropriate dose of rocuronium.
  Arms: Deep neuromuscular block
Procedure: Moderate neuromuscular block — Moderate neuromuscular block will be obtained via appropriate dose of rocuronium.
  Arms: Moderate neuromuscular block

SUMMARY:
Increased intracranial pressure (IICP) is a common problem in traumatic brain injuries and many medical diseases. Early recognition of IICP can save lives. Several invasive and non-invasive methods have been described for IICP diagnosis. In recent years, ultrasonographic measurement of optic nerve sheath diameter (ONSD) has become a popular method due to its high sensitivity and specificity for IICP estimation. Studies have shown that ONSD's ultrasonographic measurement correlates with the IICP and can detect intracranial hypertension. The ONSD measurement has advantages such as being easily applied by the clinician at the bedside, being non-invasive, providing immediate results, reproducibility and low cost. It is known that artificial carbon dioxide pneumoperitoneum created in laparoscopic surgeries increases intracranial pressure.However, it is not easy to estimate the degree of changes in ICP during laparoscopic surgery under general anesthesia. In the literature, there are many studies on the sonographic measurement of optic nerve sheath diameter to evaluate the effects of trendelenburg position on intracranial pressure with the use of different anesthetic drugs in laparoscopic surgeries. In addition, there are studies reporting that deep neuromuscular blockade in laparoscopic surgeries increases surgical vision and decreases analgesic requirement in postoperative period. The relationship between neuromuscular block level and intracranial pressure is not clear. From this point of view, the investigators would like to evaluate the effect of moderate and deep neuromuscular block level on intracranial pressure by sonographic measurement of optic nerve sheath diameter in laparoscopic cholecystectomy operations performed with standard pressure artificial carbon dioxide pneumoperitoneum.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years
* ASA I-II
* Patients undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* Intracranial hypertension
* Glaucoma
* Chronic obstructive pulmonary disease
* Pseudotumor cerebri
* Cerebral venous sinus thrombosis
* İntraoperative hemodynamic instability
* Mean arterial blood pressure<65 mmHg
* Body mass index> 35
* Asthma
* Kidney or liver problems
* Lupus
* Crohn's disease or ulcerative colitis
* Previously had any gastrointestinal bleeding
* Hypertension
* Peripheral arterial disease
* Angina, heart attacks, or mild or moderate heart failure
* Stroke

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | During surgery
  Sonographic optic nerve sheath measurements will be made 5 times, preoperatively, 5 minutes after endotracheal intubation, 5 minutes after pneumoperitoneum, 5 minutes after pneumoperitoneum is terminated and after extubation

SECONDARY OUTCOMES:
Headache | 24 hours
  The severity of the headache in the first 24 hours postoperatively(0=never, 1= rarely, 2= sometimes, 3= very often, 4= always)
Postoperative nausea and vomiting score | 24 hours
  Nausea-vomiting were assessed with postoperative nausea and vomiting scale (PONV) (0=no PONV, 1= mild nausea, 2= severe nausea or vomiting once, 3= vomiting more than once)
Patient satisfaction score | 24 hours
  Patient satisfaction measured using a NRS 1 to 10 (1 = unsatisfied; 10 =very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Yeşiltaş, Instructor, Principal Investigator — BEZMİALEM VAKIF UNIVERSITY